CLINICAL TRIAL: NCT03692728
Title: Increased Risk of Attention Deficit Hyperactivity Disorder Among Children With Bilateral Congenital Cataracts
Brief Title: Increased Risk of ADHD Among Children With Bilateral Congenital Cataracts
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Prof., Sun Yat-sen University
Other Study IDs: CCPMOH2018- China9
Record Dates: First submitted 2018-09-29; First posted 2018-10-02 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-09

CONDITIONS: Childhood Cataract
Keywords: congenital cataract; attention deficit hyperactivity disorder; Conners'Parent Rating Scale-48
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CC children: CC children were registered members of the Childhood Cataract Program of the Chinese Ministry of Health (CCPMOH). All of them were diagnosed with CC by two experienced pediatric ophthalmologists based on a comprehensive evaluation of the onset age (within one year after birth), morphological features of lens opacity, family history, and detailed medical records.
  Interventions: Other: Psychological and Behavioral Problems
- NV children: NV children were recruited from the Optometry Department of the ZOC as the control group. NV was defined as BCVA ≥0.3 (log MAR) in children between 3-5 years old or BCVA ≥0.15 (log MAR) in children older than 5 years. Children with strabismus and high refractive error (myopia or hyperopia: >6.0 Diopters; astigmatism: >3.0 Diopters) were excluded from NV group.
  Interventions: Other: Psychological and Behavioral Problems

INTERVENTIONS:
Other: Psychological and Behavioral Problems — Differences in age and sex between the CC and NV groups were compared using the independent samples t test and Chi-square test, respectively. Comparisons of abnormal rates between the CC and NV groups were performed using the Chi-square test. Scores on all subscales recorded for the CC group were compared with those of the NV group and the Chinese urban norm using the independent samples t test and one-sample t test, respectively.

SUMMARY:
In this study, the investigators conducted a cross-sectional, face-to-face investigation to evaluate the behavioral and psychological disorders and the risk of ADHD among children with bilateral congenital cataracts using the Conners'Parent Rating Scale (CPRS) questionnaire, an assessment tool for screening ADHD that obtains parental reports of childhood behavioral problems in research and clinical settings.15-17 Age-matched children with normal vision and the Chinese urban norm were used as controls.

ELIGIBILITY:
Inclusion Criteria:

* CC children and NV children aged 3-8 years presenting to the Zhognshan Ophthalmic Center between July and December 2016.

Exclusion Criteria:

* Patients complicated with systemic manifestations, such as Lowe syndrome, Marfan syndrome, and Down syndrome, were excluded.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: hospital-based
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Risk of ADHD | 2016.7-12
  The Conners' Parent Rating Scale 48 (CPRS-48) contains 5 evaluating subscales, including the conduct problems, learning problems, psychosomatic, impulsiveness/hyperactivity, and anxiety subscales. A total of 48 items are included in the questionnaire, and each item is scored from 0 to 3 (0 represents the best, 3 represents the worst). The final scores of the 5 subscales are defined as the mean scores of the corresponding items: conduct problems (2+8+14+19+20+21+22+23+27+33+34+39)/12; learning problems (10+25+31+37)/4; psychosomatic (32+41+43+44+48)/5; impulsiveness/hyperactivity (4+5+11+13)/4; anxiety (12+16+24+47)/4; and the hyperactivity index (4+7+11+13+14+25+31+33+37+38)/10. Final scores and the five subscales of the CPRS-48 between two groups were compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China